CLINICAL TRIAL: NCT03301272
Title: Effectiveness of Onabotulinumtoxin A on Reduction of Rest Tremor in Parkinson's Disease: a Pilot Study
Brief Title: Effectiveness of Botox on Reducing Rest Tremor in Parkinson's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 15-1831
Record Dates: First submitted 2017-09-13; First posted 2017-10-04 (Actual); Results first posted 2020-08-17 (Actual); Last update posted 2020-08-17 (Actual); Status verified 2019-08

CONDITIONS: Parkinson Disease
Keywords: Parkinson, Botox, Tremor
MeSH Terms: conditions — Parkinson Disease; Tremor | interventions — Botulinum Toxins, Type A; Saline Solution

STUDY DESIGN:
Intervention Model Description: The study will comprise of a double blinded, crossover study where the subjects will serve as their own controls. There will be no medication changes made to Parkinson's disease medications throughout the subjects' participation in the study.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double-blinded study whereby the subject, the movement disorder specialist injecting neurotoxin, and the movement disorder specialist rating the patient will be unaware of the solution injected and/or planned for injection same day. To ensure that the injecting specialist is blinded to the solution, syringes will be premixed by a separate member of the research team and de-identified of any possible labels that would indicate the properties of the solution being administered to the subject.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Onabotulinumtoxin A Injection, then Placebo (Experimental): Participants first receive Onabotulinumtoxin A Injection and following a 3-month washout, they receive Placebo
  Interventions: Drug: Onabotulinumtoxin A Injection; Other: Placebo
- Placebo, then Onabotulinumtoxin A Injection (Experimental): Participants first receive placebo injection and following a 3-month washout, they receive Onabotulinumtoxin A Injection.
  Interventions: Drug: Onabotulinumtoxin A Injection; Other: Placebo

INTERVENTIONS:
Drug: Onabotulinumtoxin A Injection — Reconstituted 10 units/0.1 mL. Administered intramuscular once
  Other Names: Botox
Other: Placebo — 0.9% normal saline solution, mimicking Botox injection paradigm. Administered intramuscular once.
  Other Names: Normal saline

SUMMARY:
Purpose: Rest tremor in Parkinson's disease is notoriously difficult to treat through pharmacological measures, currently only predictably attenuated by the invasive deep brain stimulation surgery. The investigators hope to find some predictable and clinically meaningful attenuation of tremor with targeted use of onabotulinum toxin on muscles involved in creating the tremor.

Participants: 16 subjects who meet United Kingdom (UK) brain bank criteria for Parkinson's disease with medically refractory rest tremor of at least 3 cm amplitude.

Procedures (methods): Subjects will be blinded to receive either sham saline injection versus onabotulinum toxin injections directed to muscle groups felt to be clinically involved in causing the oscillatory movement of the tremor. Assessment of tremor severity and functional improvement from baseline after injection will occur within group (i.e. each subject will serve as their own control).

Hypotheses:

1. (A) Onabotulinumtoxin A significantly attenuates the amplitude of medically-refractory rest tremor of the upper limb in Parkinson's patients as compared to sham injections; as measured by reduction in the Movement Disorders Society Unified Parkinson's Disease Rating Scale (MDS-UPDRS) tremor subscore.

1. (B) Onabotulinumtoxin A significantly improves the limb function of Parkinson's patients with medically-refractory rest tremor of the upper limb as compared to sham injections; as measured by an increase in Action Research Arm Test (ARAT) scores.

DETAILED DESCRIPTION:
For purposes of properly identifying muscles intended for injection, a portable electromyography will be attached to an appropriate gauge electromyography-guided botulinum toxin needle, which in turn will be used to hear/see motor evoked potentials (MEPs). Subjects will be asked to activate the muscle while needle is inserted to ensure proper placement of the needle in the desired muscle prior to injection of study solution.

ELIGIBILITY:
Inclusion Criteria:

1. At least 45 years of age, and no more than 80 years of age.
2. Meet UK Parkinson's disease brain bank diagnostic criteria
3. Have clinical evidence of rest tremor of one or both upper extremities defined as involuntary, rhythmic oscillations about any joint within the upper extremities
4. Rest tremor amplitude must be at minimum 3 cm as determined by expert opinion by a movement disorders specialist. Confirmation of amplitude measurement will be obtained from the Px1 prior to active participation in the study but will not be used for inclusion/exclusion in study participation.
5. Rest tremor must be historically refractory to at least 2 categories of medications typically used as anti-parkinsonian agents including levodopa formulations, dopamine agonists, amantadine, and anticholinergics.
6. Participants must be able to make no changes to their anti-parkinsonian medications for 150 days (study duration). Ability and safety to do so must also be determined by the participant's treating physician and confirmed in writing prior to participating.
7. Able to provide informed consent

Exclusion Criteria:

1. History of having undergone botulinum toxin injections for any other condition previously
2. Allergy to carbidopa or levodopa.
3. Prescreening Montreal Cognitive Assessment (MoCA) score less than 22
4. Prescreening muscle weakness as determined by Medical Research Council grade less than 5/5 on direct testing in the upper limb afflicted with rest tremor.
5. Pregnancy: documentation of non-pregnancy by urine pregnancy test will be obtained from all women of child-bearing potential prior to participation
6. Infection at the proposed injection site
7. Those with a pre-existing, concomitant neuromuscular disorder
8. Compromised respiratory function
9. History of having undergone deep brain stimulation surgery for any condition

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2018-03-22 (Actual); Primary Completion 2019-08-21 (Actual); Study Completion 2019-08-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel A Roque, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- UNC Hospitals Neurology Clinic, Chapel Hill, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- OnabotulinumtoxinA Injection, Then Placebo: Participants first receive OnabotulinumtoxinA Injection and following a 3-month washout, they receive Placebo
  OnabotulinumtoxinA Injection: Reconstituted 10 units/0.1 mL. Administered intramuscular once
  Placebo: 0.9% normal saline solution, mimicking Botox injection paradigm. Administered intramuscular once.
- Placebo, Then OnabotulinumtoxinA Injection: Participants first receive placebo injection and following a 3-month washout, they receive Onabotulinumtoxin A Injection.
  OnabotulinumtoxinA Injection: Reconstituted 10 units/0.1 mL. Administered intramuscular once
  Placebo: 0.9% normal saline solution, mimicking Botox injection paradigm. Administered intramuscular once.
Period: First Intervention (30 Days)
Arm/Group | OnabotulinumtoxinA Injection, Then Placebo | Placebo, Then OnabotulinumtoxinA Injection
Started | 7 | 9
Completed | 7 | 9
Not Completed | 0 | 0
Period: Washout (90 Days From 1st Intervention)
Arm/Group | OnabotulinumtoxinA Injection, Then Placebo | Placebo, Then OnabotulinumtoxinA Injection
Started | 7 | 9
Completed | 7 | 9
Not Completed | 0 | 0
Period: Second Intervention (30 Days)
Arm/Group | OnabotulinumtoxinA Injection, Then Placebo | Placebo, Then OnabotulinumtoxinA Injection
Started | 7 | 9
Completed | 7 | 9
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Placebo, Then OnabotulinumtoxinA Injection: Participants first receive placebo injection and following a 3-month washout, they receive OnabotulinumtoxinA Injection.
  OnabotulinumtoxinA Injection: Reconstituted 10 units/0.1 mL. Administered intramuscular once
  Placebo: 0.9% normal saline solution, mimicking Botox injection paradigm. Administered intramuscular once.
- Total: Total of all reporting groups
Arm/Group | OnabotulinumtoxinA Injection, Then Placebo | Placebo, Then OnabotulinumtoxinA Injection | Total
Number analyzed (Participants) | 7 | 9 | 16
Age, Continuous [Mean (Full Range); unit: years] | 65.7 [47 to 79] | 64.7 [49 to 77] | 65.5 [47 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 5 | 8 | 13
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 7 | 9 | 16
Chosen Limb for Study [Count of Participants; unit: Participants]
  Right Arm | 4 | 5 | 9
  Left Arm | 3 | 4 | 7
Mean Number of Parkinson's Medications Failed Prior to Enrollment [Mean (Standard Deviation); unit: Failed Medications] | 3.29 (1.25) | 3.0 (1.22) | 3.13 (1.20)
Levodopa Equivalent Dosing (LED) [Mean (Standard Deviation); unit: mg] — Levodopa Equivalent Dosing (LED) gives a rough way to compare two Parkinson's medications. All medications for Parkinson's can be compared in level of effect to Levodopa, the most consistently used medication for this disease.
  mg | 98.29 (54.10) | 162.22 (103.53) | 134.25 (89.22)

OUTCOME MEASURES:

1. Primary Outcome: Change in the MDS-UPDRS Tremor Subscore
Description: The Movement Disorders Society Unified Parkinson's Disease Rating Scale (MDS-UPDRS) is a clinimetric assessment of subjective and objective symptoms and signs of Parkinson's disease created by the Movement Disorder Society. MDS-UPDRS retains the four-scale structure with a reorganization of the various subscales. The subscale used in this study is Part III's tremor subscore (3.17). The subscale has a 0-4 rating, where 0 = normal, 1 = slight, 2 = mild, 3 = moderate, and 4 = severe. Higher MDS-UPDRS scores reflect worse tremor/motor function. Larger differences will infer greater effect size for the intervention. Score drops over time imply improvement in tremor/motor function.
Time Frame: Prior to onabotulinumtoxinA injection and at 30 days after injection
Population: One participant was unavailable to complete assessment during defined window.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Groups:
- OnabotulinumtoxinA Injection: Participants receive OnabotulinumtoxinA Injection.
  OnabotulinumtoxinA Injection: Reconstituted 10 units/0.1 mL. Administered intramuscular once
- Placebo: Participants receive placebo injection.
  Placebo: 0.9% normal saline solution, mimicking Botox injection paradigm. Administered intramuscular once.
Arm/Group | OnabotulinumtoxinA Injection | Placebo
Number analyzed (Participants) | 16 | 15
score on a scale | 0.25 [-0.246 to 0.746] | 0.27 [-0.342 to 0.876]
Statistical Analysis 1: Comparison: OnabotulinumtoxinA Injection vs Placebo; Test type: Other; p = 0.5, Regression, Linear — The threshold for statistical significance is 0.05; Difference in differences = 0

2. Secondary Outcome: Change in the ARAT Score
Description: The Action Research Arm Test (ARAT) is an evaluated measure to assess specific changes in limb function after neurologic sequelae. It assesses a person's ability to handle objects differing in size, weight and shape and therefore can be considered to be an arm-specific measure of activity limitation. The ARAT is a 19 item measure divided into 4 sub-tests (grasp, grip, pinch, and gross arm movement). Performance on each item is rated on a 4-point ordinal scale: 3: Performs test normally 2: Completes test, but takes abnormally long or has great difficulty 1: Performs test partially 0: Can perform no part of test. The maximum score on the ARAT is 57 points (possible range 0 to 57). Higher ARAT scores reflect greater preservation of function in tested arm. Larger differences will infer greater effect sizes for the intervention. Score drops over time imply worsening limb function.
Time Frame: Prior to onabotulinumtoxinA injection and at 30 days after injection
Population: Two participants were unavailable to complete assessments during defined window.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | OnabotulinumtoxinA Injection | Placebo
Number analyzed (Participants) | 15 | 15
score on a scale | 53.67 [49.06 to 58.27] | 55.47 [54.30 to 56.63]

3. Secondary Outcome: Correlation Between MDS-UPDRS Tremor Subscore and Px1 Tremor Amplitude
Description: MDS-UPDRS retains the four-scale structure with a reorganization of the various subscales. The subscale used is Part III's tremor subscore 3.17. The subscale has a 0-4 rating: (0=no tremor, 1=<1cm, 2=1-3 cm, 3=3-10 cm, 4=>10cm). Higher scores reflect worse tremor amplitude. Larger differences infer greater effect size. The Px1 is a novel, external measuring device using motion-capture technology to determine the frequency, direction and amplitude of movement between hand joints. Movement is captured without ever applying direct pressure on the limb. Output includes tremor frequency in Hz and distance traveled by a hand joint as compared to other joints on the hand in cm. The largest tremor amplitude measured by Px1 was acquired 3x/visit, values averaged then compared with the amplitude range corresponding to MDS-UPDRS tremor subscore. This process was repeated for all subjects for Visits 1-4 comparing all values using Spearman correlation coefficient.
Time Frame: At Visit 1, prior to 1st injection through Visit 4, 30 days after last injection
Measure: Number; unit: Spearman Correlation Coefficient
Arm/Group | OnabotulinumtoxinA Injection | Placebo
Number analyzed (Participants) | 16 | 16
Spearman Correlation Coefficient | 0.6225 | 0.4354

4. Secondary Outcome: Change in Tremor Amplitude in Centimeters (cm) as Measured by Px1
Description: The Px1 is a novel, external measuring device which uses motion-capture technology to determine the frequency, direction, and amplitude of movement between joints within the hand. Oscillatory movement is captured using a camera system and without ever applying any direct pressure upon the limb. Output includes tremor frequency in (Hertz Hz), and distance traveled by a hand joint as compared to other joints on the hand in centimeters (cm)
Time Frame: Prior to onabotulinumtoxinA injection and at 30 days after injection
Population: Given that the Px1 tool was simultaneously undergoing validation during the trial, using the tool to determine the differences in tremor amplitude was deemed inappropriate.
Arm/Group | OnabotulinumtoxinA Injection | Placebo
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Change in Tremor Frequency in Hertz (Hz) as Measured by Px1
Description: as for outcome 4
Time Frame: Prior to onabotulinumtoxinA injection and at 30 days after injection
Population: Given that the Px1 tool was simultaneously undergoing validation during the trial, using the tool to determine the differences in tremor frequency was deemed inappropriate.
Arm/Group | OnabotulinumtoxinA Injection | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were included starting with the Screening Visit up to and including Visit 5, a total of approximately 150 days.
Groups:
- Onabotulinumtoxin A Injection: Participants receive Onabotulinumtoxin A Injection.
  OnabotulinumtoxinA Injection: Reconstituted 10 units/0.1 mL. Administered intramuscular once
Arm/Group | Onabotulinumtoxin A Injection | Placebo
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 6/16 | 2/16
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Onabotulinumtoxin A Injection (N=16) | Placebo (N=16)
Weakness of Injected Limb (Musculoskeletal and connective tissue disorders) | 5 (5) | 2 (2)
Pain of Injected Limb (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-12-03): https://cdn.clinicaltrials.gov/large-docs/72/NCT03301272/Prot_SAP_000.pdf